CLINICAL TRIAL: NCT05649150
Title: The Influence of Physical Activity Level on Lumbar Movement Control and Standing Balance in Adults With and Without Low Back Pain.
Brief Title: Influence of Physical Activity Level on Lumbar Movement Control
Status: Completed | Type: Observational
Sponsor: National Cheng Kung University (Other)
Responsible Party: Principal Investigator, YI-JU TSAI, Professor, National Cheng Kung University
Other Study IDs: NCKU-2022
Record Dates: First submitted 2022-11-23; First posted 2022-12-13 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Low Back Pain
Keywords: Physical activity; Lumbar movement control; Motor control exercise; Standing balance; Proprioception
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy group: For healthy group A.K.As adults without LBP are: (1) aged from 20 to 65 years old, (2) no specific low back pain in the past 6 months.
- LBP group: The inclusion criteria for adults with LBP are: (1) aged from 20 to 65 years old, (2) persistent LBP for more than 3 months.

SUMMARY:
This study aims to compare the two groups of low back pain and health adults. To investigate the relationship among lumbar movement control, standing balance and physical activity. Methods used in the study will be clinical tools such as proprioception test, lumbar movement control, timed one-leg- standing balance and Y-balance test according to the Mat.

DETAILED DESCRIPTION:
Low back pain (LBP) is a leading cause of disability that results in significant health and socioeconomic problems. Most of the LBP is non-specific and altered motor control is one of the possible causes. Motor control exercise (MCE) thus has been recently developed as a non-operative intervention for LBP. Recently, a series of lumbar movement control (LMC) tests have been advocated to evaluate impaired motor control of lumbar. To perform a coordinated movement pattern, normal proprioception (part of neural system) is thought to be essential. Poor proprioception related to delayed muscle response and altered motor control which possibly leading to deficits in postural control and balance in LBP population. Study showed standing balance was related to higher physical activity (PA) which has been promoted in all adults and proper amount is at least 150 to 300 minutes of moderate-intensity aerobic physical activity; or at least 75 to 150 minutes of vigorous-intensity aerobic physical activity per week for substantial health benefits. As we know, there is no specific research about the relationship among PA, LMC and standing balance. Therefore, the purposes of the study are to investigate (1) the influence of different level of PA on LMC tests; (2) the influence of PA on standing balance; (3) the relationship of battery of LMC tests and standing balance in adults with and without LBP.

It is expected to recruit total 160 participants with and without LBP. The inclusion criteria for adults with LBP are: (1) aged from 20 to 65 years old, (2) persistent LBP for more than 3 months. For adults without LBP are: (1) aged from 20 to 65 years old, (2) no specific low back pain in the past 6 months. All the participants will fill in International PA Questionnaire (IPAQ), Short form Taiwan Version, perform proprioception test for the lumbar spine, LMC tests, timed one-leg standing balance, and Y-balance test for the lower quarter (YBT-LQ). After finishing the examination, all the data will be analyzed by mix analysis of variance (ANOVA) and Chi-square analysis. Bonferroni post-hoc tests will be used to identify the significance within each analysis. Level of statistical significance was set at p<0.05.

Keywords: Physical activity, motor control exercise, lumbar movement control, standing balance, proprioception

ELIGIBILITY:
Inclusion Criteria:

* For adults with LBP are: (1) aged from 20 to 65 years old, (2) persistent LBP for more than 3 months.
* For adults without LBP are: (1) aged from 20 to 65 years old, (2) no specific low back pain in the past 6 months.

Exclusion Criteria: (for both groups)

* Musculoskeletal symptoms of lower extremity in the past 6 months
* History of surgeries, fractures, or ruptures to the musculoskeletal structures on the lower limbs and spine
* Congenital spinal pathologies and deformities
* Sensory and neurological deficits
* Pregnancy
* Body mass indexes (BMI) >30 kg/m2
* Self-reported symptoms of dizziness
* Visual, vestibular or balance problems
* Other conditions affecting balance (eg, drug or alcohol consumption)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Health adults and adults with LBP
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Lumbar proprioception (joint repositioning error of lumbar spine) | One day
  Joint repositioning error of lumbar spine will be measured by the difference between starting to the finishing position. Five trials will be tested and the average of the difference will be recored for analysis.
Lumbar movement control ability | One day
  Lumbar motor control is a self-made battery according to the previous studies. The lumbar movement control tests included 10 items. And the passed number of tests will be recorded for analysis.
One-leg standing balance | One day
  Timed balance tests will be exanimated for static one-leg standing balance in four conditions. The subjects will be instructed to one leg standing in barefoot, arm folded across the chest, on solid surface or foam surface with eyes opened and closed. 3 trial for each conditions and the average of the 3 trials will be recored into analysis
Dynamic standing balance | One day
  Y-balance test- lower quarter (YBT-LQ) will be used for assessing dynamic standing balance. Participants stand on one leg in the center of the YBT-LQ and reaching the gesture leg into three different directions (anterior, posterio-lateral, posterior-medial). The reaching distance will be recored in centimeters. Three for each direction, the average will be normalized by leg length and be recorded into analysis.
Oswestry Disability Index | One day
  Oswestry Disability Index is a self-reported questionnaire for assessing disability of LBP group. The sum score of the Oswestry Disability Index will transformed into percentage for analysis.
International PA Questionnaire (IPAQ) | One day
  IPAQ is a self-reported questionnaire for assessing physical activity. The total MET-mins/week will be recorded for analysis.
Fear-Avoidance Beliefs Questionnaire (FABQ) | One day
  FABQ is an self-reported questionnaire for assessing the fear-avoidance in low back pain group. The sum of the score of the 16 questions will be transformed into percentage for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ju Tsai, Study Chair — National Cheng Kung University
Locations (1):
- National Cheng Kung University, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided